CLINICAL TRIAL: NCT03211741
Title: Longterm Efficiency and Safety of Intravitreal Injections With Bevacizumab in Patients With Neovascularisation or Macular Edema
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EudraCT number: 2013-005056-15
Record Dates: First submitted 2017-06-12; First posted 2017-07-07 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-12

CONDITIONS: Retinal Neovascularization; Macular Edema
Keywords: Bevacizumab
MeSH Terms: conditions — Retinal Neovascularization; Macular Edema | interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- open label (Other)
  Interventions: Drug: Bevacizumab Injection [Avastin]

INTERVENTIONS:
Drug: Bevacizumab Injection [Avastin] — Bevacizumab 1.25mg/0.05 mL will be injected intravitreally using one 30-gauge x 1/2-inch injection needle vials are for single eye use only.

SUMMARY:
Although the safety and efficacy of bevacizumab has been established in several phase 3 trials, there is only little documented about the long-term safety and efficacy in the 'real-world practice' in large populations from different regions.

Therefore the investigators evaluate the long-term safety and efficacy of intravitreal treatment with bevacizumab by registration of best corrected visual acuity, side-effects and central retinal thickness as measured with the ocular coherence tomography if available. This will allow the investigators to compare the results of their centre with the results of several phase 3 trials from the literature and will guide improvements in their treatment protocols.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years of either gender
2. Written informed consent must be obtained before any intravitreal injection of bevacizumab is performed
3. Visual impairment predominantly due to abnormal new vessel ingrowth and/or macular edema. The presence of fluid (intraretinal, subretinal or sub-RPE) detected clinically or on the ocular coherence tomography.

If both eyes are eligible for the study, both eyes can be included in the study.

Exclusion Criteria:

1. Women who are pregnant or breastfeeding (pregnancy defined as the state of a female after conception until the termination of gestation, confirmed by a positive human chorionic gonadotropin laboratory test (> 5mIU/mL)
2. Women of child bearing potential must be practicing effective contraception implemented during the trial and for at least 28 days following the last dose of study medication
3. Tromboembolic event (CVA or transient ischemic attack, AMI) less than 3 months prior to the intravitreal injection of bevacizumab
4. History of hypersensitivity for bevacizumab.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2013-11-22 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Best Corrected Visual Acuity | every visit, up to ten years
  will be performed with a 1, 3 or 6 month interval (or more frequent) as long as there are signs of disease activity
Slit lamp examination | every visit, up to ten years
  will be performed with a 1, 3 or 6 month interval (or more frequent) as long as there are signs of disease activity
Dilated Fundoscopy | every visit, up to ten years
  will be performed with a 1, 3 or 6 month interval (or more frequent) as long as there are signs of disease activity
Central Retinal Thickness | annually, up to ten years
  central retinal thickness as measured with the ocular coherence tomography
Fluorescein Angiography and Ocular Coherence Tomography | annually, up to ten years
  fluorescein angiography and ocular coherence tomography. The necessity of these investigations is determined by the degree of activity and as deemed necessary by the investigator.

SECONDARY OUTCOMES:
side-effects | annually, up to ten years

CONTACTS AND LOCATIONS:
Locations (1):
- Ghent University Hospital, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No